CLINICAL TRIAL: NCT02864797
Title: Health Related Quality of Life of Patients With Gynecologic Cancers: Feasibility Study of a Prospective and Pragmatic Cohort
Brief Title: Feasibility Study of a Prospective and Pragmatic Cohort
Acronym: GYNEQOL-Pilot
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Centre Hospitalier Universitaire de Besancon (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: P/2014/238
Record Dates: First submitted 2016-07-29; First posted 2016-08-12 (Estimated); Last update posted 2017-10-13 (Actual); Status verified 2017-10

CONDITIONS: Gynecologic Cancers
Keywords: Health related quality of life; patient reported outcomes; cohort; e-health

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Health related quality of life collected via CHES (Experimental): Health related quality of life (QoL) is collected at each follow-up visit using tablets computer and CHES software.
  Interventions: Other: Health related quality of life collected via CHES

INTERVENTIONS:
Other: Health related quality of life collected via CHES — Health related quality of life (QoL) is collected at each follow-up visit using tablets computer and CHES software. Thus, QoL's results are directly presented to clinicians via the CHES, in order to be considered as part of the supportive care strategy at the end of the study

SUMMARY:
Gynecologic cancers (cancers of cervix, endometrium, ovary, vagina, and vulva) represent an important part of the female cancer in France with more than 15 000 new cases in 2012. As considerable progress have been made in diagnostic and therapeutic strategies, an important part of the gynecologic cancers are diagnosed at an early stage and globally, the after treatment overall survival rate is estimated to more than 80% at five years. Thus, it is of evident interest to study health related Quality of Life (QoL) among these patients who will continue to live after their cancer and to consider QoL as a primary end-point, beyond overall survival.

The GYNEQOL (health related Quality Of Life of women with GYNEcologic cancer) group is a working group initiated in Besançon and whose goal is to investigate QoL of gynecologic cancers' patients. It gathers several entities from the hospital of Besançon, namely the Methodology and Quality of Life in Oncology Unit, the Gynecologic Unit and the Oncology Unit. The GYNEQOL study is a project of a prospective cohort study, in a pragmatic clinical practice, with the main objective of longitudinally collecting and analyzing QoL data of these women.

The pilot phase, GYNEQOL-Pilot, restricted to the hospital of Besançon, has started in September 2015 with the goal of assessing the feasibility of the cohort. The feature of this study is that patients answer to QoL questionnaires using tablets computer and the Computer-based Health Evaluation System software (CHES). Indeed, use of electronic solutions to collect patient reported outcomes is drastically increasing those last years. It has been underlined that routinely collecting symptoms could increase both QoL and survival among cancer patients. It enables to use these data in real-time in routine practice by presenting QoL scores to physicians in simple graphical histograms for both transversal and longitudinal measurements and it ensures a reliable data collection.

DETAILED DESCRIPTION:
Gynecologic cancers (cancers of cervix, endometrium, ovary, vagina, and vulva) represent an important part of the female cancer in France with more than 15 000 new cases in 2012. As considerable progress have been made in diagnostic and therapeutic strategies, an important part of the gynecologic cancers are diagnosed at an early stage and globally, the after treatment overall survival rate is estimated to more than 80% at five years. Thus, it is of evident interest to study health related Quality of Life (QoL) among these patients who will continue to live after their cancer and to consider QoL as a primary end-point, beyond overall survival.

The GYNEQOL (health related Quality Of Life of women with GYNEcologic cancer) group is a working group initiated in Besançon and whose goal is to investigate QoL of gynecologic cancers' patients. It gathers several entities from the hospital of Besançon, namely the Methodology and Quality of Life in Oncology Unit, the Gynecologic Unit and the Oncology Unit. The GYNEQOL study is a project of a prospective cohort study, in a pragmatic clinical practice, with the main objective of longitudinally collecting and analyzing QoL data of these women.

The pilot phase, GYNEQOL-Pilot, restricted to the hospital of Besançon, has started in September 2015 with the goal of assessing the feasibility of the cohort. The feature of this study is that patients answer to QoL questionnaires using tablets computer and the Computer-based Health Evaluation System software (CHES). Indeed, use of electronic solutions to collect patient reported outcomes is drastically increasing those last years. It has been underlined that routinely collecting symptoms could increase both QoL and survival among cancer patients. It enables to use these data in real-time in routine practice by presenting QoL scores to physicians in simple graphical histograms for both transversal and longitudinal measurements and it ensures a reliable data collection.

Objectives The main objective is to collect and analyse QoL of gynecologic cancer patients in a prospective and pragmatic cohort study.

The primary endpoint will be QoL assessed by the European Organization for Research and Treatment of Cancer (EORTC) QLQ-C30 (Core Quality of Life Questionnaire), for the following targeted dimensions : global health, emotional, social and functional roles and fatigue

The secondary objectives are to assess those endpoints :

* the participation rate
* the acceptability of the use of the CHES and tablets computer
* use of the QoL results by the physicians
* occurence and type of missing data
* attrition

Study population All adult patients with gynecologic cancers (ovarian, endometrial and cervical cancers), treated in the University hospital of Besançon, and who gave their informed consent, are prospectively included. Patients who do not well understand French, who have cognitive impairment or who do not have social insurance are not included.

Data collection Socio-demographic, socio-economic (occupational group, attained education, income), behavioural (physical activity), previous history and familial history of cancer, clinical, medical data, biomarkers, therapeutic strategies, toxicities and QoL will be prospectively collected at inclusion and throughout the follow-up. As we are in the context of pragmatic clinical practice, visits are based on the usual follow-up of gynecologic cancer patients.

QoL will be assessed using EORCT QLQ-C30 questionnaire and the specific modules QLQ-CX24 (cervix), QLQ-OV28 (ovaries) and QLQ-EN24 (endometrium), using a time-driven design. These auto-questionnaires will be administrated with the CHES and the help of an clinical research associate at inclusion, before treatment, 3 weeks after treatment and at each "routine" follow-up visit during at least 6 months. If patients do not want to use tablet computer, "pen-paper questionnaire" will be administered.

Statistical analyses Usual statistical methods will be used for description of socio-demographic, socio-professional, clinical of patients at inclusion and of QoL throughout the follow-up. Those characteristics will be described considering cancer localizations and stages and used therapeutics/surgeries. We will also described the participation rate.

The acceptability of the use of the CHES and tablets computer and the use of the QoL results by the physicians will be qualitatively described.

Missing data will be described by assessing profile of patients with missing data, occurence of missing data for each QoL item, incomplete QoL questionnaire rate and type of missing data (missing at random, missing completely at random, missing not at random).

ELIGIBILITY:
Inclusion Criteria:

* patient with newly diagnosed gynecologic cancer (ovaries, endometrium, cervix, vagina, vulva, fallopian tube), whatever the stage and histological type.
* patient treated at Besançon University Hospital
* patient aged of 18 years old or older
* patient who do understand French
* patient without any major cognitive impairment
* patient who hav signed the informed consent
* patient affiliated to the French social insurance

Exclusion Criteria:

* patient with recurrent cancer
* patient with legal incapacity or limited legal capacity
* patient without any social insurance
* patient unlikely to cooperate

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 116 (Actual)
Dates: Start 2015-09-29 (Actual); Primary Completion 2018-08-22 (Estimated); Study Completion 2018-08-22 (Estimated)

PRIMARY OUTCOMES:
Health related quality of life (QoL) | month 18
  The primary endpoint will be QoL assessed by the EORTC QLQ-C30, for the following targeted dimensions : global health, emotional, social and functional roles and fatigue

SECONDARY OUTCOMES:
Participation rate | at the last inclusion, up to 12 months
  the rate of number of included patients on number of eligible patients
acceptability of the use of the CHES and tablets computer | at study completion, up to 24 months
  How did patients perceived the use of tablets computer and CHES software, qualitative assessment by the clinical research associates
frequency of use of the QoL results by the physicians | at study completion, up to 24 months
  how many times physicians used the CHES in their clinical practice.
occurence and type of missing data | at study completion, up to 24 months
  count of QoL missing data at each time point
attrition | at study completion, up to 24 months
  count of patients lost of follow up at study completion

CONTACTS AND LOCATIONS:
Overall Officials: Rajeev RAMANAH, MD PhD, Principal Investigator — CHU Besançon; Elsa KALBACHER, MD, Principal Investigator — CHU Besançon
Locations (1):
- CHU Besançon, Besançon, France

IPD SHARING:
Plan to Share IPD: No